CLINICAL TRIAL: NCT00702793
Title: Safety and Tolerability of Varenicline When Used for Smoking Cessation/Reduction in Individuals With Severe and Persistent Mental Illness: An Open Label Pilot Trial
Brief Title: Safety and Tolerability of Varenicline in Schizophrenia (SATOVA)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of British Columbia (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Ric Procyshyn, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H07-02939
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Schizoaffective; Psychosis
Keywords: Smoking cessation; schizophrenia; schizoaffective; psychosis; varenicline; champix; chantix; nicotine dependence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking Cessation; Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Smoking cessation drug - varenicline
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 0.5 mg/d for days 1 to 3, 0.5 mg twice daily for days 4 to 7, then 1 mg twice daily through week 12. Administration of twice daily dosing should be at least 8 hours apart.
  Other Names: Champix; Chantix

SUMMARY:
This is a 15 week trial to determine (1) the safety and tolerability of varenicline when used for smoking cessation/reduction in individuals with schizophrenia; (2) if treatment with varenicline affects the symptoms of schizophrenia.

DETAILED DESCRIPTION:
Researchers are looking to recruit a total of 50 subjects at Riverview and Forensic Psychiatric Hospitals who would like to reduce or quit smoking cigarettes. This open label pilot study will gather information regarding the safety and tolerability of varenicline in subjects who have been diagnosed with schizophrenia or schizoaffective disorder. Consenting subjects will be prescribed varenicline as follows: varenicline 0.5 mg/d for days 1 to 3, 0.5 mg twice daily for days 4 to 7, then 1 mg twice daily through week 12. The research team will meet with the subject once a week for twelve weeks and the subject will be interviewed and asked to complete questionnaires about his/her psychiatric symptoms, tobacco use and nicotine dependence. The measures used include the FTND, PANSS, CGI-I, CGI-S, ESRS, UKU, BARS, WSWS, QSU-brief, mCEQ, and the OAS-M. The CGI-SS will also be completed throughout the study as well as once weekly for three weeks following the completion of the study (Post-Study follow-up visits 1-3).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with a diagnosis of schizophrenia or schizoaffective disorder
* Individuals between the ages of 19 and 65 years of age
* Individuals that had smoked 10 cigarette/day or more during the previous year, and had no period of smoking abstinence longer than 3 months in the past year
* Individuals that are not expected to be discharged from hospital within 4 months.

Exclusion Criteria:

* Clinically significant allergic reactions to the study medication
* Clinically significant abnormalities in the screening laboratory values
* Subjects at significant risk of self-harm
* Previous treatment with varenicline
* Women who are pregnant, breast-feeding, or of child-bearing potential not using adequate contraception
* Men not using adequate contraception
* Use of medications that might interfere with the study medication evaluation

  * Nicotine replacement
  * Nortriptyline
  * Clonidine

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in the symptoms of the primary illness. These outcomes will be measured at study visits 1, 2, 4, 8, and 12. | 12 weeks

SECONDARY OUTCOMES:
Safety and tolerability, nicotine dependence, and smoking cessation/reduction. These outcomes will be measured at study visits 1-12. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ric M. Procyshyn, Ph.D, Principal Investigator — University of British Columbia; Alasdair Barr, Ph.D, Study Director — University of British Columbia; Joyce Coutts, MD, Study Director — Forensic Psychiatric Institute; Sean Flynn, MD, Study Director — University of British Columbia; Chris Schenk, MD, Study Director — Riverview Hospital; William Honer, MD, Study Director — University of British Columbia